CLINICAL TRIAL: NCT01692704
Title: Downstaging of Unresectable Intrahepatic or Hilar Cholangiocellular Carcinoma by Selective Intra-arterial Floxuridine and Systemic Cisplatin and Gemcitabine. A Dose Finding Single Center Phase IIa Study
Brief Title: Downsizing of Unresectable Cholangiocarcinoma by Combined Intravenous and Intra-arterial Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONK-USZ-003
Record Dates: First submitted 2012-06-06; First posted 2012-09-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Cholangiocellular Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAI with FUDR & systemic cisplatin and gemcitabin (Experimental): FUDR: 0.2mg/kg/day continuously i.a. for 14 days Cisplatin: 25mg/m2 i.v. Gemcitabin: different doses according to dose level 600, 800, or 1000 mg/m2 i.v.
  Interventions: Drug: Selective intra-arterial floxuridine and systemic gemcitabine and cisplatin

INTERVENTIONS:
Drug: Selective intra-arterial floxuridine and systemic gemcitabine and cisplatin — Intra-arterial floxuridine:0.2 mg/KG/day for 14 days, repeated day 29. Overall 3 applications.
  Systemic cisplatin: 25 mg/m2 at days 1 and 8, repeated day 22. Overall 8 applications.
  Systemic gemcitabine: Three different dose levels will be tested; 600 mg/m2, 800 mg/m2, or 1000 mg/m2, at days 1 and 8, repeated day 22. Overall 8 applications.

SUMMARY:
An open label, prospective, non-randomized single arm study. Combination of two treatment modalities - HAI with FUDR and systemic chemotherapy with cisplatin and gemcitabine.

Definition of the maximum tolerated dose (MTD) of intravenous gemcitabine in combination with intravenous cisplatin and intra-arterial FUDR. Definition of safety and toxicity of this combined regional and systemic treatment approach. Definition of the response rate after 3 months of hepatic intra-arterial chemotherapy with continuous infusion FUDR with or without ligation of the right or left portal vein, in combination with 3 months of systemic cisplatin and gemcitabine in patients with unresectable intrahepatic or hilar CCC.

A total of 9-18 patients are required. 3-6 patients per dose level. A maximum of three dose levels (1 - 3) has been defined.

Statistical Methodology: Traditional 3+3 dosing algorithm to find MTD.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically proven cholangiocellular carcinoma including gallbladder cancer.
* Non-resectable cholangiocellular carcinoma as judged within an interdisciplinary tumor-board including senior hepatobiliary surgeons. Non- resectability is based on insufficient remnant liver volume.
* Patient is not a candidate for liver transplantation
* WHO Performance Score 0 or 1
* No extrahepatic tumor, as evaluated by PET/CT scan of the chest and the abdomen/pelvis with the exception of potentially resectable small lung nodules or hilar lymph node involvement.
* The assessment is done within 21 days before registration.
* Adequate liver function or kidney function tests, including any of the following:

  * Bilirubin < 2 x ULN
  * Aspartate-Aminotransferase (AST) < 5 x ULN
  * Alanine-Aminotransferase (ALT) < 5 x ULN
  * Alkaline phosphatase < 5 x ULN
  * Estimated creatinine clearance > 60 ml/min (using the Cockcroft formula)
* Adequate hematological values:

  * Hemoglobin > 80 G/L
  * Leucocytes > 3.00 G/L,
  * Neutrophils > 1.00 G/Ll
  * Platelets > 100 G/L
* Signed written informed consent
* Patient age >/= 18 years
* Presentation of the case at the interdisciplinary tumor-board attended by hepatobiliary surgeons, oncologists, hepatologists and radiologists
* Women who are not breastfeeding and are using effective contraception if sexually active, who are not pregnant and agree not to become pregnant during the 12 months thereafter. A negative pregnancy test before inclusion into the trial is required for women < 50 years.
* Men who agree not to father a child during participation in the trial or during the 12 months thereafter.
* Patient compliance and geographic proximity allow proper staging and follow- up.

Exclusion criteria:

* Anatomic variant in arteriogram which prevents selective delivery of the chemotherapy to the liver
* Life expectancy < 3 months
* Severe medical or psychiatric co-morbidity prohibiting the planned treatment or the giving of informed consent
* Any man or woman of childbearing age in case of inadequate contraception
* Pregnancy or breastfeeding woman
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
* Treatment in clinical trial within 30 days prior to trial entry.
* Active heart disease defined as congestive heart failure > NYHA class 2
* Past or current history (within the last 2 years prior to treatment start) of other malignancies except basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Inability or unwillingness to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) of intravenous gemcitabine with concomitant administration of FUDR-HAI and intravenous cisplatin. | 6 weeks
  Dose limiting toxicities will be assessed to define the maximum tolerated dose (MTD) of gemcitabine in combination with fixed doses of cisplatin and FUDR. DLTs are per protocol prespecified AE or laboratory abnormalities observed during the first 6 weeks of study treatment. The MTD is one dose level below the dose level that caused DLTs in ≥ one third of patients (2 or more in a cohort of 6 patients), as determined by a traditional 3+3 algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Samaras, MD, Principal Investigator — University Hospital Zurich, Department of Oncology
Locations (1):
- University Hospital Zurich, Department of Oncology, Zurich, Canton of Zurich, Switzerland